CLINICAL TRIAL: NCT03289260
Title: Adjuvant Imiquimod Therapy to Reduce Recurrence Rate in Patients After Surgical Therapy of Anal HPV (Human Papilloma Virus)-Lesions
Brief Title: Adjuvant Anal Imiquimod Therapy in Anal HPV-lesions: AdAM-trial
Acronym: AdAM
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, Irmgard E Kronberger, MD, Leading Consultent, Medical University Innsbruck
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AdAM_2017
Record Dates: First submitted 2017-09-19; First posted 2017-09-20 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Anogenital Human Papillomavirus Infection; Condyloma Anal
Keywords: Condylomata acuminata, Fulguration, Imiquimod
MeSH Terms: conditions — Condylomata Acuminata | interventions — Imiquimod; Diathermy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional Arm (Experimental): Imiquimod 5% cream therapy Fulguration
  Interventions: Drug: Imiquimod 5% cream; Procedure: Fulguration
- Placebo Arm (Placebo Comparator): Placebo cream therapy Fulguration
  Interventions: Drug: Placebo cream; Procedure: Fulguration

INTERVENTIONS:
Drug: Imiquimod 5% cream — Patients receive topical Imiquimod therapy for 12 weeks.
  Other Names: Aldara
  Arms: Interventional Arm
Drug: Placebo cream — Patients receive topical Doritin therapy for 12 weeks
  Other Names: Doritin
  Arms: Placebo Arm
Procedure: Fulguration — Surgical Excision and Fulguration of condyloma

SUMMARY:
AdAM is a prospective, randomized, controlled, double-blinded, monocentric trial in patients receiving surgical therapy due to anal HPV infection.

Aim of the study is to evaluate efficacy of combination therapy (surgical therapy + topical Imiquimod-therapy). It is planned to include 200 patients.

100 patients receive surgical therapy+ topical Imiquimod therapy, 100 patients receive surgical therapy + topical Placebo therapy

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and willingness to sign and date a written consent document
* Male and female patients >= 18 years of age
* Negative urine/serum pregnancy test
* Indication for surgical therapy of anal HPV lesions

Exclusion Criteria:

* Participation in another clinical study with experimental therapy
* Diagnosis and therapy of HPV associated lesions in the last 12 months
* Known intolerance of hypersensitivity to Imiquimod
* Women who are pregnant of lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-11-15 (Estimated); Primary Completion 2024-11-15 (Estimated); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
Difference in recurrence rates between the two arms | 12 months
  Recurrence is evaluated by clinical examination (proctoscopy)

SECONDARY OUTCOMES:
CD4 (cluster of differentiation 4) cell count | 12 months
  Influence of CD4 cell count in the subgroup of HIV positive patients

CONTACTS AND LOCATIONS:
Overall Officials: Dietmar Öfner-Velano, MD, Study Director — University Hospital for Visceral, Transplant and Thoracic Surgery
Locations (1):
- Visceral-, Transplant- and Thoracic Surgery, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: Undecided